CLINICAL TRIAL: NCT03438903
Title: Comparison of Repeatability Between Swept-source and Spectral-domain Optical Coherence Tomography for Measuring Inner Retinal Thickness in Various Retinal Diseases
Brief Title: Comparison of Repeatability Between SS and SD-OCT for Measuring Retinal Thickness in Various Retinal Diseases
Status: Completed | Type: Observational
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yong Un shin, Assistant professor, Hanyang University
Other Study IDs: 2017-10-013
Record Dates: First submitted 2018-02-12; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Macula Abnormality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal group: Healthy subjects without any ocular problems Repeat exams of OCT device (SD and SS-OCT)
  Interventions: Device: Repeat exams of OCT device
- Retinal diseases group: Patients with various macular diseases Repeat exams of OCT device (SD and SS-OCT)
  Interventions: Device: Repeat exams of OCT device

INTERVENTIONS:
Device: Repeat exams of OCT device — All 2 consecutive OCT examinations were performed by 1 experienced technician, in the order of SD-OCT and SS-OCT. The interval was 10 minutes between examinations by each OCT devices

SUMMARY:
Comparison of intradevice repeatability of thickness measurements for macular area in the eyes with normal and various retinal diseases using SS-OCT and SD-OCT

DETAILED DESCRIPTION:
The investigators studied the intradevice repeatability of thickness measurements for total retina, retinal nerve fiber layer (RNFL) and ganglion cell-inner plexiform (GC-IPL) layers of macular area in the eyes with normal and various retinal diseases using SS-OCT and SD-OCT and compared the repeatability between two devices.

ELIGIBILITY:
Inclusion Criteria:

* Age-matched normal group was composed of subjects with age over at least 19 years,
* a best-corrected visual acuity of 20/25 or higher,
* normal fundus and intraocular pressure (IOP) < 21mm Hg.

Exclusion Criteria:

* an spherical equivalent (SE) larger than ± 6 D,
* cataract graded as more severe than grade 3 (Lens Opacities Classification System III),
* a history of glaucoma and optic nerve diseases, or a history of vitrectomy.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal control : 36 eyes of 36 subjects
  retinal disease group: 78 eyes of 78 patients
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
To compare repeatability between swept-source optical coherence tomography (SS-OCT) and spectral-domain OCT (SD-OCT) devices for the measurement of retinal thickness in various retinal diseases. | Each device was examined twice consecutively within one minutes. After one OCT device exam, another OCT exam was performed immediately. The interval between test devices did not exceed 5 minutes.
  Comparison of Intraclass correlation coefficient (ICC) and coefficients of variability (CV) between devices

SECONDARY OUTCOMES:
To compare repeatability according to the degree of macular thickness | Each device was examined twice consecutively within one minutes. After one OCT device exam, another OCT exam was performed immediately. The interval between test devices did not exceed 5 minutes.
  To compare the repeatability of retinal thickness according to central macular thickness in eyes with retinal diseases

CONTACTS AND LOCATIONS:
Overall Officials: Mincheol Seong, MD, PhD, Study Chair — Hanyang University
Locations (1):
- Hanyang University Guri Hospital, Guri-si, Gyeonggi-do, South Korea